CLINICAL TRIAL: NCT00629304
Title: Multicenter Assessment of the PDA-FIT System in Type 1 Diabetic Patients With Chronic Failure of Intensive Insulin Therapy and Conventional Care. The TELEDIAB-1 STUDY
Brief Title: Multicenter Assessment of the PDA-FIT System in Type 1 Diabetic Patients
Acronym: TELEDIAB-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DCIC 07 08
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2009-08

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; PDA phone (Personal Digital Assistant); HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Placebo Comparator): standard visit at 3 and 6 months
  Interventions: Device: placebo
- 2 (Active Comparator): PDA-FIT system + standard visit at 3 and 6 months
  Interventions: Device: VISITS + PDA-FIT system
- 3 (Active Comparator): PDA-FIT system + 12 telephone visits + standard visit at 6 months
  Interventions: Device: PDA-FIT System + telephone follow-up

INTERVENTIONS:
Device: placebo — Patients will have face to face visits at 3 and 6 months and no PDA-FIT system. Patients will record glycemia on paper support.
  Other Names: paper support for glycemia; face to face visits at 3 and 6 months; without PDA-FIT system
  Arms: 1
Device: VISITS + PDA-FIT system — patients will have face to face visits at 3 and 6 months + PDA-FIT system
  Other Names: face to face visits at 3 and 6 months; PDA-FIT system
  Arms: 2
Device: PDA-FIT System + telephone follow-up — patients will received PDA-FIT system + a telephone follow up (12 phone calls) and a face to face visit at 6 months
  Other Names: face to face visit at 6 months; telephone visits each 2 weeks; PDA-FIT system
  Arms: 3

SUMMARY:
TELEDIAB-1 is a national, multicenter, controlled, randomised trial. The Primary objective of the TELEDIAB-1 study is to demonstrate that the PDA-FIT system (PDA-Phone and/or telemonitoring) is able to improve metabolic control of chronically uncontrolled type 1 diabetic patients, despite intensive insulin therapy (multiple daily injections with basal-bolus insulin or insulin pump), as compared with conventional care.

Main judgment criteria: comparison of HbA1c means between the 3 groups at 6 months

DETAILED DESCRIPTION:
Secondary Objectives :

1. To assess the improvement of blood glucose control and quality of life in patients using the PDA-FIT system
2. To assess the improvement in diabetes care provided by the use of the PDA-FIT system
3. Satisfaction of patients and physicians towards the PDA-FIT system

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes mellitus for ≥ 12 months or more (including C-peptide negative secondary diabetes)
* age > 18 y.o.
* intensive insulin basal-bolus therapy for ≥ 6 months. At inclusion, patients should be treated, either with a combination of a basal, long-acting insulin and insulin rapid analog before each meal, or with rapid insulin analog delivered with a pump
* chronically uncontrolled diabetes with HbA1c ≥ 8 % during the past 12 months and at inclusion

Exclusion Criteria:

* patient with unstable associated evolutive pathology
* patient who need a more frequent diabetic follow up (than in the protocol)
* patient with a education teaching within the 3 months before inclusion
* patient with a hemoglobinopathy
* patient with toxicomania, alcoholism or psychological troubles
* type 2 diabetes patients
* patient who don't need strict metabolic objectives
* pregnant or parturient women
* person with no freedom (prisoner)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-09; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Comparison of HbA1c mean between the 3 groups | at 6 months

SECONDARY OUTCOMES:
Absolute HbA1c differences (M0-M6) | inclusion and M6
HbA1c changes at M0, M3 and M6 | inclusion, M3 and M6
Percentage of patients reaching HbA1c <7.5% at 6 months | 6 months
Mean of blood glucose values as provided by glucose meters during the 14 days prior to inclusion and prior to the 6 months-visit | 14 days prior to inclusion and prior to M6
Frequency of severe hypoglycaemic episodes and ketoacidosis episodes during the study period | study period
Frequency of symptomatic benign hypoglycaemic episodes during the week prior to inclusion and prior to the 6 months-visit | week before inclusion and prior to M6
8-point blood glucose profiles at inclusion and 6 months | inclusion and M6
Quality of life at inclusion and 6 months, using the DHP scale and the Satisfaction item of the DQOL questionnaire | inclusion and M6
Improvement in diabetes care, as assessed by the change in blood glucose testing frequency, reflected by the glucose meter memory | study period
Time spent by physicians with patients during visits (either face to face visits or phone call visits) and time spent by patients during transport, waiting time and lost working time | study period
Satisfaction of patients and physicians with the system and willingness to carry on the use of the system in routine care | 6 months
Effective number of patients carrying on the use of the system in routine care, at their own expense and in agreement with their physician | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Yves BENHAMOU, MD PHD, Study Chair — University Hospital, Grenoble
Locations (18):
- France (18):
  - Centre Hospitalier de Belfort Montbéliard, Belfort, Belfort
  - CHU Jean Minjoz, Besançon, Besancon
  - CH SUD Francilien, Corbeil-Essonnes, Corbeil Essonnes
  - University Hospital Grenoble, Grenoble, Grenoble
  - CHRU Lille, Lille, Lille
  - Hopital Edouard Herriot, Lyon, Lyon
  - CHU Marseille Hôpitaux Sud, Marseille, Marseille
  - Chu Montpellier, Montpellier, Montpellier
  - CHU Hôpital Jeanne d'Arc, Nancy, Nancy
  - CHU Nantes, Nantes, Nantes
  - Hopital Hotel Dieu, Paris, Paris
  - Hopital COCHIN, Paris, Paris
  - HOPITAL Saint Louis, Paris, Paris
  - Hopital Haut Leveque, Pessac, Pessac
  - CHU Rennes, Rennes, Rennes
  - Hopital Bellevue, Saint-Etienne, Saint Etienne
  - Centre Hospitalier Strasbourg, Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse, Toulouse

REFERENCES:
- [Derived] Charpentier G, Benhamou PY, Dardari D, Clergeot A, Franc S, Schaepelynck-Belicar P, Catargi B, Melki V, Chaillous L, Farret A, Bosson JL, Penfornis A; TeleDiab Study Group. The Diabeo software enabling individualized insulin dose adjustments combined with telemedicine support improves HbA1c in poorly controlled type 1 diabetic patients: a 6-month, randomized, open-label, parallel-group, multicenter trial (TeleDiab 1 Study). Diabetes Care. 2011 Mar;34(3):533-9. doi: 10.2337/dc10-1259. Epub 2011 Jan 25. PMID 21266648